CLINICAL TRIAL: NCT00870766
Title: Computer Tomography (CT) Trial of Acute Abdomen
Acronym: PRACTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Pekka Miettinen, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH5200617
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Acute Abdomen
MeSH Terms: conditions — Abdomen, Acute

ARMS (2):
- CT (Active Comparator): All patients in the CT arm undergo abdominal CT scanning within 24 hours of admission to the ER.
  Interventions: Procedure: Abdominal contrast-enhanced CT scanning
- Current practice (No Intervention): The patients in the current practice arm are referred to radiological examinations, such as US, plain radiography or CT, based on the clinical need only.

INTERVENTIONS:
Procedure: Abdominal contrast-enhanced CT scanning — Contrast-enhanced (iohexol 350 mgI/ml, 100 ml IV) CT scanning
  Arms: CT

SUMMARY:
The purpose of this study is to determine the impact of routinely performed early CT scanning in terms of diagnostic accuracy, patient management and cost-effectiveness compared to current imaging practice in patients suffering from acute abdomen.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* abdominal pain > 2h and < 7 days

Exclusion Criteria:

* pregnancy
* acute abdominal trauma
* allergy to iodinated contrast media
* severe renal insufficiency
* metformin medication combined with elevated plasma creatinin level
* lack of cooperation (if informed consent is not possible)
* abdominal pain combined with bleeding shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | at discharge and/or 2-3 mo follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland